CLINICAL TRIAL: NCT05824442
Title: Evaluation of a New Multiplex Quantitative PCR Technique for the Diagnosis of Echinococcosis
Acronym: HIS-QPCR-ECH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022/737
Record Dates: First submitted 2023-01-27; First posted 2023-04-21 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Echinococcosis; Diagnosis
Keywords: High sensitive qPCR
MeSH Terms: conditions — Echinococcosis; Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological sample (Experimental): Blood sample
  Interventions: Biological: Blood sample for multiplex QPCR technique

INTERVENTIONS:
Biological: Blood sample for multiplex QPCR technique — Blood sampling specifically for qPCR Echino at inclusion and one year after

SUMMARY:
Echinococcosis is a severe parasitosis caused by the development of the tapeworm larva Echinococcus multilocularis, responsible for alveolar echinococcosis (AE) or Echinococcus granulosus, responsible for cystic echinococcosis (CE). The treatment is based on surgery (only possible in 30 to 40% of cases) and/or on a benzimidazole antiparasitic treatment, especially albendazole. Albendazole is only parasitostatic, it slows down the development of the parasite but does not kill it. It is often prescribed for life. Monitoring the effectiveness of the treatment is therefore necessary, requiring radiological and serological monitoring once or twice a year. Being a chronic disease whose treatment is not always curative, patients quality of life is impacted, with a high level of anxiety described in some patients.

The diagnosis, evoked on radiological arguments, is then confirmed by serological techniques, whose sensitivity for EA diagnosis is good (95%) in the absence of immunosuppression (now observed in 25% of EA patients). Sensitivity is lower for CE diagnosis (70% or even less than 50% in certain clinical forms).

Quantitative real-time PCR (QPCR) techniques on blood samples are now used in many infectious pathologies to quantify the circulating DNA load, and improve diagnosis and therapeutic monitoring. The presence of circulating parasitic DNA has been reported in both types of echinococcosis.

A new Echinococcus spp.multiplex QPCR technique (QPCR-Echino) allowing the detection of DNA from E. multilocularis and different species of the E. granulosus complex of European occurrence, in different types of biological samples, has recently been developed in the French National Reference Center for Echinococcosis laboratory.

The investigators wish to evaluate QPCR-Echino for the detection of DNA in tissues, as well as in blood, for the diagnosis of Echinococcosis. This technique could improve the sensitivity of biological diagnosis, especially in immunocompromised patients, who often experience significant diagnostic delays, and could also provide information on the virulence and viability of the strains involved.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged >18 years with a diagnosis of echinococcosis (Alveolar Echinococcosis or Cystic Echinococcosis) established according to the reference criteria
* Signature of the informed consent form indicating that the subject has understood the purpose and the procedures required by the study and that he agrees to participate in the study and to comply with the requirements and restrictions about this study
* Affiliation to a French social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate in the study and/or low cooperation anticipated by the investigator
* Subject without health insurance
* Pregnant woman
* Subject being in the period of exclusion from another study or provided by the "national volunteer file".

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Performance indicators of a new diagnosis technique based on multiplex quantitative PCR | 1 year
  sensitivity of DNA detection by QPCR-Echino in tissues (operating specimens, biopsies, puncture fluids) and in blood (plasma)

CONTACTS AND LOCATIONS:
Overall Officials: Delphine VERHOEVEN-WEIL, MD, Principal Investigator — CHU Besançon
Locations (1):
- MILLON, Besançon, France

IPD SHARING:
Plan to Share IPD: No